CLINICAL TRIAL: NCT01968668
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Safety and Efficacy of Different Oral Doses of BAY94-8862 in Japanese Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Nephropathy
Brief Title: Safety and Efficacy of Different Oral Doses of BAY94-8862 in Japanese Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Nephropathy (ARTS-DN Japan)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16816
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Nephropathies
Keywords: BAY94-8862; MR antagonist; Diabetic nephropathy; Japanese patients
MeSH Terms: conditions — Diabetic Nephropathies | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- BAY94-8862 (1.25 mg) (Experimental)
  Interventions: Drug: BAY94-8862
- BAY94-8862 (2.5 mg) (Experimental)
  Interventions: Drug: BAY94-8862
- BAY94-8862 (5 mg ) (Experimental)
  Interventions: Drug: BAY94-8862
- BAY94-8862 (7.5 mg) (Experimental)
  Interventions: Drug: BAY94-8862
- BAY94-8862 (10 mg) (Experimental)
  Interventions: Drug: BAY94-8862
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BAY 94-8862 (15 mg) (Experimental)
  Interventions: Drug: BAY 94-8862
- BAY 94-8862 (20 mg) (Experimental)
  Interventions: Drug: BAY 94-8862

INTERVENTIONS:
Drug: BAY94-8862 — 1.25 mg BAY94-8862 tablet once daily in the morning
  Arms: BAY94-8862 (1.25 mg)
Drug: BAY94-8862 — 2.5 mg BAY94-8862 tablet once daily in the morning
  Arms: BAY94-8862 (2.5 mg)
Drug: BAY94-8862 — 5 mg BAY94-8862 tablet once daily in the morning
  Arms: BAY94-8862 (5 mg )
Drug: BAY94-8862 — 7.5 mg BAY94-8862 tablet once daily in the morning
  Arms: BAY94-8862 (7.5 mg)
Drug: BAY94-8862 — 10 mg BAY94-8862 tablet once daily in the morning
  Arms: BAY94-8862 (10 mg)
Drug: Placebo — Placebo tablet once daily in the morning
  Arms: Placebo
Drug: BAY 94-8862 — 15 mg BAY 94-8862 tablet once daily in the morning
  Arms: BAY 94-8862 (15 mg)
Drug: BAY 94-8862 — 20 mg BAY 94-8862 tablet once daily in the morning
  Arms: BAY 94-8862 (20 mg)

SUMMARY:
This study will be conducted in Japanese subjects with type 2 diabetes mellitus and the clinical diagnosis of Diabetic Nephropathy( DN) using a multi-center, randomized, adaptive, double-blind, placebo-controlled, parallel-group design.

Primary objective of the study is investigate the change of Urinary Albumin to Creatine Ratio (UACR) after treatment with different oral doses of BAY94-8862 given once daily from baseline to Visit 8 (Day 90)

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects with type 2 diabetes mellitus and a clinical diagnosis of DN (Diabetic Nephropathy) treated with at least the minimal recommended dose of an Angiotensin Converting Enzyme Inhibitor (ACEI) and/or Angiotensin Receptor Blocker (ARB)
* Subjects with a clinical diagnosis of Diabetic Nephropathy (DN) based on at least 1 of the following criteria:

  * Persistent very high albuminuria defined as Urinary Albumin to Creatine Ratio (UACR) of >/=300 mg/g (>/=34 mg/mmol) in 2 out of 3 first morning void samples and estimated glomerular filtration rate (eGFR) >/=30 mL/min/1.73 m2 but <90 mL/min/1.73 m2 Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) or
  * Persistent high albuminuria defined as UACR of >/=30 mg/g but <300 mg/g (>/=3.4 mg/mmol but <34 mg/mmol) in 2 out of 3 first morning void samples and eGFR>/=30 mL/min/1.73 m2 but <90 mL/min/1.73 m2 (CKD-EPI)
* Serum potassium </=4.8 mmol/L at both the run-in visit and the screening visit

Exclusion Criteria:

* Non-diabetic renal disease (confirmed by biopsy)
* Known bilateral clinically relevant renal artery stenosis (>75%)
* Glycated hemoglobin(HbA1c) >12% at the run-in visit or the screening visit
* UACR >3000 mg/g (339 mg/mmol) in any of the urinary first morning void samples at the run-in visit or screening visit
* Hypertension with mean sitting systolic blood pressure (SBP) >/=180 mmHg or mean sitting diastolic blood pressure (DBP) >/=110 mmHg at the run-in visit or mean sitting SBP >/=160 mmHg or mean sitting DBP >/=100 mmHg at the screening visit
* Subjects with a clinical diagnosis of heart failure with reduced ejection fraction (HFrEF) and persistent symptoms (New York Heart Association class II-IV) at the run-in visit
* Concomitant therapy with eplerenone, spironolactone, any renin inhibitor, or potassium-sparing diuretic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2014-10-09 (Actual); Study Completion 2014-11-07 (Actual)

PRIMARY OUTCOMES:
Change of urinary albumin-to creatinine ratio | Baseline and 90 days

SECONDARY OUTCOMES:
Change in serum potassium concentration | Baseline and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Japan (14):
  - Nagoya, Aichi-ken
  - Saijō, Ehime
  - Kurume, Fukuoka
  - Obihiro, Hokkaido
  - Amagasaki, Hyōgo
  - Koga, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Kahoku-gun, Ishikawa-ken
  - Sakaidechō, Kagawa-ken
  - Izumisano, Osaka
  - Yao, Osaka
  - Katsushika-ku, Tokyo
  - Osaka

REFERENCES:
- [Derived] Snelder N, Heinig R, Drenth HJ, Joseph A, Kolkhof P, Lippert J, Garmann D, Ploeger B, Eissing T. Population Pharmacokinetic and Exposure-Response Analysis of Finerenone: Insights Based on Phase IIb Data and Simulations to Support Dose Selection for Pivotal Trials in Type 2 Diabetes with Chronic Kidney Disease. Clin Pharmacokinet. 2020 Mar;59(3):359-370. doi: 10.1007/s40262-019-00820-x. PMID 31583611
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/